CLINICAL TRIAL: NCT04235582
Title: Encouraging Opioid Abstinence Behavior: Incentivizing Inputs and Outcomes - Pilot
Brief Title: Incentives to Decrease Opioid Use - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Chicago (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1095
Record Dates: First submitted 2019-11-20; First posted 2020-01-22 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2021-01

CONDITIONS: Substance-Related Disorders; Opioid-Related Disorders; Behavior Therapy
Keywords: opioid-use disorder; substance-use disorder; addiction; contingency management; dynamicare
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Behavior, Addictive | interventions — Amyloid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Outcomes Group (Experimental): During the intervention period, the "Outcomes" group will receive incentives for abstaining from drug use. Patients in this group will receive the same services and urine drug-test schedule as standard of care and a similar mobile app and debit card as the Inputs group. However, the app will prompt patients in this group to submit saliva drug tests through their mobile phones on a random schedule (averaging three tests per week). Patients will receive immediate financial rewards in exchange for submitting drug-negative samples. Saliva tests typically have a window of detection between 24-48 hr after drug use.
  Interventions: Behavioral: App + Outcomes Contingency Management
- Inputs Group (Experimental): Will receive incentives for behaviors that are inputs to abstaining from drug use. Patients in this group will receive the same services and urine drug-test schedule as standard of care. Additionally, patients will be registered for a mobile phone app provided by DynamiCare Health and provided with a linked debit card. The app will prompt patients to complete actions that are inputs to abstinence an average of three times per week. These actions will be tailored to the patient's individual needs, and may include:
  * Drug adherence to prescribed SUD pharmacotherapy
  * Attendance at individual and group psychotherapy sessions
  Interventions: Behavioral: App + Inputs Contingency Management
- Combination Group (Experimental): Will receive interventions from both Inputs and Outputs groups, as well as standard of care therapy services and urine drug tests an average of three times per week, total. Interventions include incentives for:
  * Drug adherence to prescribed SUD pharmacotherapy
  * Attendance at individual and group psychotherapy sessions
  * Random saliva tests
  Interventions: Behavioral: App + Inputs Contingency Management; Behavioral: App + Outcomes Contingency Management

INTERVENTIONS:
Behavioral: App + Inputs Contingency Management — The app has programmed contingencies whereby incentives can be earned for behaviors that are inputs to abstaining from drug use (e.g., attending psychotherapy or taking SUD psychopharmacology).
  Arms: Combination Group; Inputs Group
Behavioral: App + Outcomes Contingency Management — The app has programmed contingencies whereby incentives can be earned for outcomes of abstaining from drug use (e.g., drug-negative saliva samples on saliva opioid tests).
  Arms: Combination Group; Outcomes Group

SUMMARY:
The purpose of this study is to address two key questions in the literature on incentives for substance use. The first question is whether it is more effective to directly incentivize the outcome of interest - drug abstinence - or to incentivize behaviors that are inputs into the production of abstinence. This study will compare two versions of the incentive program: one that incentivizes inputs to achieving abstinence and one that incentivizes the outcome of abstinence. The second question is how to optimize the size of incentives over time to maximize incentive effectiveness. This will be done by randomly varying the size and timing of incentives offered to participants in both the Inputs and Outcomes groups. The incentive amounts will then be varied across participants and time to fit a structural model of abstinence behaviors over time. The model will be used to describe the optimal shape of incentives over time.

DETAILED DESCRIPTION:
Numerous studies have tested whether providing incentives to encourage abstinence from drugs can further reduce drug abuse in a drug-treatment setting. The results are promising: Incentives to reduce opioid abuse increase the average duration of abstinence by 25 - 60% relative to medication and counseling alone. Similar effects have been demonstrated repeatedly across a wealth of populations, substance-abuse disorders, and payment methodologies.

Despite evidence that incentives are effective and the increasing need for effective approaches to combat the addiction crisis, incentive programs have not been widely implemented. A key barrier is that while the benefits are largely borne by patients and taxpayers, there are large logistical costs that must be borne by clinics: most existing incentive programs involve manual, in-person measurement of behaviors, and prize or voucher purchase and delivery by clinic staff. The significant clinic-level legwork necessary to set up these programs, including setting up behavioral and payment tracking systems, training staff, etc., have prevented the programs from scaling widely. In sum, prior experience has consistently shown that incentives increase duration of treatment and decrease substance abuse, but the logistical complications remain a hurdle to implementation.

This will be the first randomized evaluation of an innovative, scalable incentives program for opioid addiction delivered through a mobile application. The application, which was developed by our implementing partner, DynamiCare Health, provides a "turnkey" solution that health clinics can easily prescribe. The app enables remote monitoring of behavior; for example, drug tests can be administered in patients' homes, as patients submit "selfie-videos" showing them taking saliva drug tests, which are then verified by trained remote staff. Treatment adherence can similarly be checked through GPS tracking for on-site methadone pharmacotherapy. The efficacy of this approach has not been tested rigorously before.

This study will address two key knowledge gaps in the logistics of existing incentive program design for opioid addiction. First, the first technology t for remote monitoring of abstinence behavior for opioid use will be tested. Remote monitoring of abstinence from cigarettes and alcohol has been integral in reducing the costs and extending the potential reach of incentive programs for people with nicotine/tobacco and alcohol use disorders (e.g. to vulnerable or rural populations), and this study promises to do the same for opioid addiction. The second gap is in remote delivery of incentives. After a behavior is verified, the app will deliver incentives to patients as cash available on a linked debit card. The delay between monitoring of the target behavior and the delivery of financial incentives has been shown to be a significant moderator of treatment effect size. This technology allows patients to receive incentives almost immediately following the undertaking of the incentivized behavior: a first in incentives for opioid addiction.

Another novel feature of this design is that can allow assessment of a gap in the literature on incentive delivery: comparing both the isolated effects of incentives and of the monitoring needed to implement an incentive program. In addition to a control group, this study includes both monitoring groups and incentives groups. While existing literature on incentives for addiction has included either a monitoring group or a control group, this is the first to include both, such that a comparison can be made between incentives that are distal (inputs) and proximal (outcome) to the targeted abstinence behavior.

Finally, this study will directly address two key open questions in the literature on incentives for drug-users. The first question is whether it is more effective to directly incentivize the outcome of interest - drug abstinence - or to incentivize behaviors that are inputs into the production of abstinence. Similarly designed studies did not detect different effects on abstinence from incentivizing treatment attendance and incentivizing cocaine abstinence among cocaine users (both were effective): however, not only was this study for a different substance use disorder, but because of differential rates of test submission among these two groups, the results were not conclusive. This study will similarly compare two versions of the incentive program: one that incentivizes inputs to achieving abstinence, and one that incentivizes the outcome of abstinence. To address differential test submission rates, the impacts of the intervention will be measured via urine drug-tests administered identically to patients in both treatments.

The second question is how to optimize the size of incentives over time to maximize incentive effectiveness. This will be assessed by randomly varying the size and timing of incentives offered to participants in both the Inputs and Outcomes groups. The variation in incentive amounts across participants and time to fit a structural model of abstinence behaviors over time. The model will be used to describe the optimal shape of incentives over time.

The results of this intervention will be directly relevant for potential users of this or similar mobile applications for incentive provision among people with opioid-use disorders, including insurers, treatment facilities, and governments.

ELIGIBILITY:
Inclusion

1. Age at least 18 years old;
2. Meet DSM-5 opioid use disorder criteria as evidenced by an opioid disorder CPT code F11 (opioid related disorders);
3. Have access to a smartphone (iOS or Android) with data plan and willing to download DynamiCare app;
4. Are in day (PHP) or partial day (IOP) AODA treatment in Aurora Health's Behavioral Health Program;
5. Are currently prescribed or will be prescribed within 1-4 days oral buprenorphine for their OUD;
6. Are likely to be helped by contingency management because at least ONE of the following conditions is true:

   1. Were first enrolled in day or partial day opioid treatment no longer than 1 week prior to providing informed consent.
   2. Currently using non-medical opioids.
   3. Regularly missing scheduled AODA appointments.
7. Understands English.

Exclusion Criteria:

1. Have evidence of active (non-substance related) psychosis that might impair participation as determined by the PI.
2. Has significant cognitive impairment that might confound participation as determined by the PI or are so significantly cognitively impaired that they have a legal guardian.

Note that pregnant women are not excluded from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fendrich, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - University of California - Santa Cruz, Berkeley, California
  - University of Chicago, Chicago, Illinois
  - Aurora Psychiatric Hospital, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benishek LA, Dugosh KL, Kirby KC, Matejkowski J, Clements NT, Seymour BL, Festinger DS. Prize-based contingency management for the treatment of substance abusers: a meta-analysis. Addiction. 2014 Sep;109(9):1426-36. doi: 10.1111/add.12589. Epub 2014 May 23. PMID 24750232
- [Background] Kurti AN, Davis DR, Redner R, Jarvis BP, Zvorsky I, Keith DR, Bolivar HA, White TJ, Rippberger P, Markesich C, Atwood G, Higgins ST. A Review of the Literature on Remote Monitoring Technology in Incentive-Based Interventions for Health-Related Behavior Change. Transl Issues Psychol Sci. 2016 Jun;2(2):128-152. doi: 10.1037/tps0000067. PMID 27777964
- [Background] Lussier JP, Heil SH, Mongeon JA, Badger GJ, Higgins ST. A meta-analysis of voucher-based reinforcement therapy for substance use disorders. Addiction. 2006 Feb;101(2):192-203. doi: 10.1111/j.1360-0443.2006.01311.x. PMID 16445548
- [Background] Petry NM, Alessi SM, Carroll KM, Hanson T, MacKinnon S, Rounsaville B, Sierra S. Contingency management treatments: Reinforcing abstinence versus adherence with goal-related activities. J Consult Clin Psychol. 2006 Jun;74(3):592-601. doi: 10.1037/0022-006X.74.3.592. PMID 16822115
- [Background] Schottenfeld RS, Chawarski MC, Pakes JR, Pantalon MV, Carroll KM, Kosten TR. Methadone versus buprenorphine with contingency management or performance feedback for cocaine and opioid dependence. Am J Psychiatry. 2005 Feb;162(2):340-9. doi: 10.1176/appi.ajp.162.2.340. PMID 15677600

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Group: Will receive interventions from both Inputs and Outputs groups, as well as standard of care therapy services and urine drug tests an average of three times per week, total. Interventions include incentives for:
  * Drug adherence to prescribed SUD pharmacotherapy
  * Attendance at individual and group psychotherapy sessions
  * Random saliva tests
  App + Inputs Contingency Management: The app has programmed contingencies whereby incentives can be earned for behaviors that are inputs to abstaining from drug use (e.g., attending psychotherapy or taking SUD psychopharmacology).
Period: Overall Study
Arm/Group | Outcomes Group | Inputs Group | Combination Group
Started | 12 | 13 | 11
Completed | 12 | 12 | 8
Not Completed | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Inputs Group: Will receive incentives for behaviors that are inputs to abstaining from drug use. Patients in this group will receive the same services and urine drug-test schedule as standard of care. Additionally, patients will be registered for a mobile phone app provided by DynamiCare Health and provided with a linked debit card. The app will prompt patients to complete actions that are inputs to abstinence an average of three times per week. These actions will be tailored to the patient's individual needs, and may include:
  * Drug adherence to prescribed SUD pharmacotherapy
  * Attendance at individual and group psychotherapy sessions
  App + Inputs Contingency Management: The app has programmed contingencies whereby incentives can be earned for behaviors that are inputs to abstaining from drug use (e.g., attending psychotherapy or taking SUD psychopharmacology).
- Combination Group: Will receive interventions from both Inputs and Outputs groups, as well as standard of care therapy services and urine drug tests an average of three times per week, total. Interventions include incentives for:
  * Drug adherence to prescribed SUD pharmacotherapy
  * Attendance at individual and group psychotherapy sessions
  * Random saliva tests
  App + Inputs Contingency Management: The app has programmed contingencies whereby incentives can be earned for behaviors that are inputs to abstaining from drug use (e.g., attending psychotherapy or taking SUD psychopharmacology).
  App + Outcomes Contingency Management: The app has programmed contingencies whereby incentives can be earned for outcomes of abstaining from drug use (e.g., drug-negative saliva samples on saliva opioid tests).
- Total: Total of all reporting groups
Arm/Group | Outcomes Group | Inputs Group | Combination Group | Total
Number analyzed (Participants) | 12 | 12 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.6) | 34.0 (8.4) | 29.9 (8.8) | 34.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant withdrew and three did not download the app
  Participants
    Female | 3 | 3 | 4 | 10
    Male | 9 | 9 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 6
  Not Hispanic or Latino | 9 | 9 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 10 | 11 | 7 | 28
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 8 | 32
Employment [Count of Participants; unit: Participants]
  Full-Time (30+ hr/week) | 2 | 3 | 1 | 6
  Part-Time (<30 hr/week) | 0 | 1 | 0 | 1
  Unemployed | 10 | 8 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence From Opioid Use
Description: The primary endpoint is the longest period of continuous abstinence from illicit opioids, where abstinence is measured using lab-verified in-person urine-tests, saliva tests, or subject reporting (in the absence of urine testing).
Time Frame: Time = 4 weeks
Population: These were any participant who had a saliva test or urine test on file at Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Outcomes Group | Inputs Group | Combination Group
Number analyzed (Participants) | 7 | 6 | 5
Participants | 6 | 5 | 5

2. Primary Outcome: Continuous Abstinence From Opioid Use
Description: as for outcome 1
Time Frame: Time = 8 weeks
Population: These were any participant who had a saliva test or urine test on file at Week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Outcomes Group | Inputs Group | Combination Group
Number analyzed (Participants) | 6 | 6 | 4
Participants | 6 | 5 | 3

3. Primary Outcome: Opioid-negative Saliva Tests at Week 12
Description: The primary endpoint is the % of opioid-negative saliva or urine tests in each group at Week 12
Time Frame: Time = 12 weeks
Population: These were any participant who had a saliva test or urine test on file at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Outcomes Group | Inputs Group | Combination Group
Number analyzed (Participants) | 7 | 8 | 5
Participants | 6 | 5 | 3

ADVERSE EVENTS:
Time Frame: These were collected during the 12 weeks the participant had access to the intervention.
Arm/Group | Outcomes Group | Inputs Group | Combination Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/8

LIMITATIONS AND CAVEATS:
This is a pilot and feasibility study with relatively few enrollees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04235582/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04235582/ICF_001.pdf